CLINICAL TRIAL: NCT04393116
Title: Patients' Guidance With Onco-Coaching and CANKADO on Systemic Chemotherapy for Metastatic Colorectal Cancer
Acronym: POSCA
Status: Completed | Type: Observational
Sponsor: Cankado GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-17-02
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a prospective, single arm, non-interventional project to evaluate the benefit/influence of individualized patient education and guidance with a web-based e-Health platform called CANKADO on patient reported outcomes (PRO) for patients with metastatic colorectal cancer. The focus will be on patient reported outcomes (PRO), distress, Quality of Life (QoL), Global Health Status, complaints and therapy relevant decisions. All patients will be medically treated according to the standards. The experimental arm will include 40 patients. Those patients will receive one initial coaching before start of therapy. Further appointments for coaching will be scheduled depending on individual patient's need. During treatment period the patient is encouraged of joining therapy actively documenting his state of health and occurring health complaints via CANKADO to give the physician a better overview on the process of patient's health behaviour and preparing him for the next doctor-patient consultation.

ELIGIBILITY:
Inclusion Criteria:

* Minumum age of 18 years
* Patient with metastatic colorectal cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic colorectal cancer in first line treatment treated in "Gemeinschaftspraxis für Hämatologie und Onkologie Langen" or "Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg"
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Development of patients' Distress | 6 months
  Evaluated using the Screening Tool for Measuring Distress described by the Practice Guidelines in Oncology - v. 1.2005 by the National Comprehensive Cancer Network

SECONDARY OUTCOMES:
Patient's Quality of Life (QoL) | 6 months
  Evaluated using the EORTC QLQ-C30, which is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials. The five functional scales, three symptom scales, one global health status / QoL scale, and six single items are calculated according to the scording procedures defined by the QL Coordinator, Quality of Life Unit, EORTC Data Center.
Patient's global health status | 6 months
  Evaluated using the EQ visual analogue scale (EQ-VAS Scale), a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (maximum value = 100) and 'The worst health you can imagine' (minimum value = 0).

CONTACTS AND LOCATIONS:
Overall Officials: Timo Schinköthe, PhD, Study Director — Cankado GmbH
Locations (2):
- Germany (2):
  - Hämato-onkologischer Studienkreis am Klinikum Aschaffenburg, Aschaffenburg
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen